CLINICAL TRIAL: NCT06472375
Title: Multicenter Randomized Clinical Trial to Assess the Clinical Benefit of 24-hour in Hospital Observation of Syncope Patients Admitted to the Cardiac Emergency Room
Brief Title: In Hospital 24 Hour Observation of Syncope Patients
Acronym: RISC
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Frederik de Lange, principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL 81736.018.22
Record Dates: First submitted 2024-02-13; First posted 2024-06-25 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- discharge: immediate discharge with ambulant HR monitoring (investigational treatment strategy) in low- and intermediate syncope patients in the setting of cardiac emergency room
  Interventions: Diagnostic Test: holter
- admission for 24 hours with rhythmobservation: discharge after 24-hour telemetric-observation (reference treatment strategy) in low- and intermediate syncope patients in the setting of cardiac emergency room
  Interventions: Diagnostic Test: holter

INTERVENTIONS:
Diagnostic Test: holter — ambulant heart rate monitor (holter) for 24 hour.

SUMMARY:
Syncope is very common and has a broad differential diagnosis. Guidelines on syncope recommend to apply guideline based syncope algorithm (SA) to identify low- / intermediate risk syncope patients and recommend to discharge these patients. The time window when to discharge these patients is not defined in the guidelines. In current medical practice low- / intermediate risk syncope patients are either immediately discharged or discharged after 24-hour observation with telemetry (TM). There seems to be an equipoise for both treatment strategies in current medical practice for these low risk syncope patients. A randomized controlled trial to compare discharge after 24 hour observation including TM with immediate discharge has never been done on the Cardiac Emergency Room (CER).

DETAILED DESCRIPTION:
The diagnosis of syncope is a worldwide clinical dilemma. Appropriate identification of low risk vs high risk will reduce inappropriate admission for 24-hour observation with TM. The Dutch Geriatrics Society prioritized syncope management on its research agenda. This project is endorsed by the Dutch Societies of Neurology, Cardiology, Geriatrics, and Internal Medicine and results in freely accessible tutorials on an educational website: www.syncopedia.org.

A randomized clinical trial that includes guideline based SA as routine medical care in the setting of a cardiac emergency room, that compares discharge after 24-hour observation with TM (reference treatment strategy) and immediate discharge (investigational treatment strategy) for low- and intermediate syncope patients will provide new insights and improve syncope health care for these patients.

ELIGIBILITY:
Inclusion Criteria:

All patients that are assessed as low- and intermediate risk syncope, are eligible for inclusion in this trial.

The initial syncope evaluation includes:

1. Complete and thorough history taking of the syncope event and past medical history
2. Physical examination including supine and standing BP measurement and
3. 12 lead ECG.

Exclusion Criteria:

A potential patient who meets any of the following criteria will be excluded from participation in this study:

1. Those aged <18 years
2. Those in whom syncope / transient loss of consciousness co-exist with trauma or other serious condition identified in the CER (massive bleeding, pulmonary embolus) or any high-risk features upon assessment with guideline based SA
3. Those with any other conditions then syncope / transient loss of consciousness for which admission is required (including social indication for admission, etc.)
4. Contraindication for early discharge as the discretion of the responsible physician
5. Those with a learning disability
6. Those presenting with pre-syncope
7. Those who are unwilling to provide informed consent (those will be asked to be enrolled for the SYNCOPE R.I.S.C-registry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Cardiac Emergency Room with low- and intermediate risk syncope.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Supraventricular tachycardia: | 24 hour after randomization
  a) Any atrial tachycardia (sustained or non-sustained ≥ 3 consecutive complexes) b) Atrio-Ventricular Nodal Re-entry Tachycardia (AVNRT) or Atrioventricular Re-Entry Tachycardia (AVRT) c) Premature Atrial Complex (PAC): >2 doublets or >2 episodes of 3 seconds duration of bi- or trigeminy d) Atrial Fibrillation de novo
Incidence of Ventricular tachycardia: | 24 hour after randomization
  a) Any Ventricular Tachycardia (sustained/non sustained) b) Ventricular Fibrillation c) Premature Ventricular Complexes: >2 doublets or >2 episodes of 3 seconds duration of bi- or trigemini
Incidence of Conduction disorders: | 24 hour after randomization
  a) Asystole >3sec (including conversion pauses) b) New first degree AV block with PQ>300 msec c) Progression first degree AV block with 15% c) 2nd degree AV block Mobitz type I and II d) 3rd degree AV block e) Any SA block
Incidence of Other events | 24 hour after randomization
  a) Syncope recurrence b) Unexplained fall with injury c) All cause death d) Cardiovascular death

SECONDARY OUTCOMES:
Comparison of Syncope related healthcare costs | 1 month
  Health care costs will be calculated on the basis of the tariffs set by the schedule of the Dutch National Health Service.
Hospital utilization and duration of total in-hospital stay for both arms | 1 month
  Hospital utilization of both treatment strategies will be quantified by the duration of the in-hospital stay from the moment of randomization.
Proportion of additional diagnoses after both treatment strategies | 24 hour after randomization
  The analysis will be conducted at the major group level, i.e. (1) reflex syncope, (2) orthostatic hypotension, (3) cardiac syncope. Diagnostic yield is defined as the number of patients receiving a diagnosis in the patient chart and is determined at two times during this trial:
  1. After performing the guideline based syncope algorithm (before enrollment of the patient) and
  2. At 24 hours after completing each treatment strategy.
Assessment of Quality of life (EQ5D - EuroQuol 5Dimensions) | up to 1 Month
  The questionnaires include a check-list to assess health care consumption (consultations, admissions), productivity, and QoL measures. 5 dimensions for describing health states. Scores are: no, mild, moderate, severe and extreme or unable to do. (can be scored as 1-5) In the questionnaire is also an Visual Analogue Scale: overall assessment of respondent's health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Assessment of Quality of life (Short Form Health Survey 12) | up to 1 Month
  Questionnaire to asses Quality of Life. Questionnaire contains closed questions with different response options. 'Yes/no', 'never(1)-always(6)' or 'no limitation(1)-severe limitation(3)'
Assessment of Quality of life (SyncopeDailyFunctioning) | up to 1 Month
  Questionnaire to assess qyality of life in daily functioning. Questionnaire contains closed questions with different response options. 'Yes/no' or '1(negative)-8(positive)'

CONTACTS AND LOCATIONS:
Overall Officials: Frederik de Lange, MD PhD, Principal Investigator — PI
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands